CLINICAL TRIAL: NCT04922957
Title: A Phase 2b Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study, Evaluating Efficacy and Safety of Allocetra-OTS in Patients With Severe or Critical COVID-19 With Associated Acute Respiratory Distress Syndrome (ARDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: strategic reprioritization
Sponsor: Enlivex Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ENX-CL-03-002
Record Dates: First submitted 2021-06-09; First posted 2021-06-11 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2022-08

CONDITIONS: Covid19
Keywords: Cell therapy; Allocetra-OTS
MeSH Terms: conditions — COVID-19 | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Intervention Model Description: 152 patients will be allocated in a 1:1 ratio between the 2 cohorts:
  1. Placebo
  2. Single Intravenous (IV) dose of Allocetra-OTS (10x10^9 cells)
Who Masked: Participant, Investigator
Masking Description: Randomization will be in a double blinding fashion. The IP will be delivered with a cover to maintain blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Ringer's lactate solution
  Interventions: Other: Placebo
- ALLOCETRA-OTS (Experimental): Single IV dose of Allocetra-OTS containing 10x10^9 cells
  Interventions: Drug: ALLOCETRA-OTS

INTERVENTIONS:
Drug: ALLOCETRA-OTS — The product contains allogeneic donor mononuclear enriched cells in the form of a liquid suspension containing early apoptotic cells.
  Other Names: Cell based therapy; Apoptotic cells
  Arms: ALLOCETRA-OTS
Other: Placebo — Ringer's lactate solution
  Arms: Placebo

SUMMARY:
This is a Phase 2b multi-center, randomized, double-blind, placebo-controlled study evaluating the efficacy and safety of intravenous (IV) Allocetra-OTS 10x10^9 cells vs placebo (1:1) in adult hospitalized patients with severe or critical Coronavirus Disease 2019 (COVID-19) with associated acute respiratory distress syndrome (ARDS). Patients will be followed for efficacy and safety for 6 months. The trial will include periodic and ad-hoc DSMB review during the study period.

DETAILED DESCRIPTION:
This is a Phase 2b multi-center, randomized, double-blind, placebo-controlled study evaluating the efficacy and safety of intravenous (IV) Allocetra-OTS 10x10^9 cells vs placebo (1:1) in adult hospitalized patients with severe or critical Coronavirus Disease 2019 (COVID-19) with associated acute respiratory distress syndrome (ARDS).

Severe and critical COVID-19 are defined as follows:

Severe COVID-19: shortness of breath at rest, or respiratory distress, or respiratory rate (RR) ≥30 per minute, or SpO2 ≤93% on room air at sea level.

Critical COVID-19: respiratory failure, requiring at least one of the following: oxygen delivered by high-flow nasal cannula or noninvasive positive pressure ventilation.

After a patient has signed the informed consent form (ICF), and after confirmation that the patient meets all eligibility criteria, the patient will be enrolled in the study. The two subpopulations, severely ill and critically ill patients, will be randomized 1:1 into the active treatment and placebo groups via two separate randomizations schemes.

Study treatment (Investigational Product or placebo) administration will occur on Day 1 as close as possible to and no later than 48 hours from randomization. Assessments, performed on Day 1 prior to study treatment administration, will be considered as baseline assessments.

Patients will be followed for efficacy and safety through 6 months. Following study treatment administration, patients will be assessed daily for a period of 7 days. The next visits are planned to occur on Days 14, 28 and 60. A safety follow-up phone call will be scheduled to occur 6 months post study treatment. Hospitalized patients will be monitored on a daily basis until discharge or up to 60 days post study treatment administration.

Blood samples for safety assessment will be analyzed locally as per institutional guidelines.

Additional blood samples will be collected for potential exploratory analyses. Such biomarker analyses will be performed centrally as per Sponsor requirements.

Patients who drop out within the interval between the randomization and study treatment administration will be replaced to keep the originally planned sample size.

The trial will include periodic and ad-hoc Data Safety Monitoring Board (DSMB) review during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female >18 and <85 years of age.
2. Laboratory confirmation of SARS-CoV-2 infection by RT-PCR from any diagnostic sampling source.
3. Patient hospitalized due to COVID-19 within 7 days prior to enrollment, meeting the criteria for severe or critical COVID-19 as follows:

   1. Severe COVID-19 - defined as shortness of breath at rest, or respiratory distress, or RR ≥30 per minute, or SpO2≤93% on room air at sea level.
   2. Critical COVID-19 - defined as respiratory failure, requiring at least one of the following: oxygen delivered by high-flow nasal cannula or noninvasive positive pressure ventilation.
4. Patient with mild to moderate ARDS:

   1. 100< PaO2/FiO2 ≤300; based on the Berlin Definition of ARDS
   2. 148< SpO2/FiO2 ≤315; based on the Kigali modification for ARDS

      * If available, PaO2 will be obtained, otherwise, SpO2 will be used for ARDS assessment.
5. Signed written informed consent by the patient.
6. Women and men who are of childbearing potential, willing to use acceptable contraceptive measures during 4 weeks from enrollment.

Exclusion Criteria:

1. Patient on IMV/ECMO.
2. Woman who is pregnant or breastfeeding.
3. Patient with weight <50 kg or >120 kg or BMI >40 kg/m^2.
4. Patient with stage 4 or 5 chronic kidney disease or estimated glomerular filtration rate <30 mL/min.
5. Patient with an active malignant tumor (diagnosed or on active treatment for the past 6 months).
6. Patient who is participating in other concurrent interventional clinical trials or has been treated with any experimental agents within 30 days prior to enrollment.
7. Patient who based on their medical history and receipt of therapies that would suggest infection, has suspected serious, active bacterial (including a suspected clinical diagnosis of current active tuberculosis [TB] or, if known, latent TB treated for less than 4 weeks with appropriate anti-TB therapy per institutional guidelines), fungal, or viral (including, but not limited to, active HBV, HCV, or HIV/AIDS) infection.
8. Patient with known immunocompromised state or immunosuppressive medications taken for indications other than SARS-CoV-2 as follows:

   * Prednisone or equivalent to a dose >10 mg/day, methotrexate >15 mg/week, within the last 60 days. cyclophosphamide, cyclosporine A (unless as ophthalmic formulation), leflunomide/teriflunomide (unless as monotherapy), tacrolimus (unless as a topical formulation), everolimus, temsirolimus, or azathioprine, in the last 60 days;
   * Methylprednisolone, dexamethasone, cortisone, or betamethasone for more than 7 days within the last 28 days or within 5 half-lives, whichever is longer;
   * Chemotherapy in the last 3 months;
   * Mycophenolate mofetil (MMF) or sirolimus for solid organ transplant or bone marrow transplant;
   * Thalidomide within the last 72 hours.
   * Anti-tumor necrosis factor (TNF) agents, interleukin (IL)-1 receptor antagonists (IL-1-RA), CTLA-4 fusion proteins, anti-CD20, anti-CD52, anti-IL-2, anti-IL-6R, anti-IL-12/23, anti-B-cell activation factor (BAFF) or integrin inhibitor agents within the last 8 weeks.
9. Patient with known New York Heart Association (NYHA) class III and IV heart failure or unstable angina, ventricular arrhythmias, ischemic heart disease, or myocardial infarction within 6 months prior to diagnosis of COVID-19.
10. Patient with known active upper gastrointestinal (GI) tract ulceration or hepatic dysfunction including but not limited to biopsy-proven cirrhosis; end-stage cirrhosis (Child Pugh Class C); portal hypertension; episodes of past upper GI bleeding attributed to portal hypertension; or prior episodes of hepatic failure, encephalopathy, or coma.
11. Patient with known idiopathic pulmonary fibrosis.
12. Patient with chronic respiratory disease requiring home oxygen therapy on a regular basis for more than 6 hours per day.
13. Patient with known chronic obstructive pulmonary disease GOLD 4 (forced expiratory volume in one second <30% predicted).
14. Patient with any medical, psychiatric or substance abuse condition, concurrent medical therapies, or abnormal laboratory values that in the opinion of the site Investigator may influence response to study product, or interfere with the study assessments.
15. Patient with GCS <13 with verbal score <5.
16. Patient with hemoglobin <8 g/dL.
17. Patient with history of chronic liver disease, evidence of acute cholangitis or cholecystitis. Patients with at least one of the following:

    * ALT or AST >10xULN (upper limit of normal)
    * Bilirubin >5xULN
    * Combination of ALT/AST >7xULN and elevated direct bilirubin >ULN
18. Patient with known history of transfusion reactions, hemolytic anemia, or repetitive allergic reaction.
19. Patient with previous history of organ allograft or stem cell transplantation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Time (days) to improvement | 28 days
  The first day, during the period of 28 days post study treatment, when a patient reached the score of 6, 7 or 8 on the 8-point ordinal scale. If no improvement is reached by Day 28, the patient will be assigned a maximal score of 29.
  The 8-point ordinal scale of the clinical severity status scores is as follows:
  Death=1; Hospitalized, on IMV or ECMO=2; Hospitalized, on noninvasive ventilation or high-flow oxygen devices=3; Hospitalized, requiring supplemental oxygen by mask or nasal canula=4; Hospitalized, not requiring supplemental oxygen=5; Hospitalized, not requiring supplemental oxygen and not requiring ongoing inpatient medical care=6; Not hospitalized, limitations on activities=7; Not hospitalized, no limitations on activities=8.
Support by IMV/ECMO | 28 days
  If required during the period of 28 days post study treatment, a patient will be assigned the maximal score of 29.
Mortality | 28 days
  Mortality by Day 28 post study treatment administration. Deceased patients will be assigned the maximal score of 29.

SECONDARY OUTCOMES:
Time (days) to improvement, defined as the first day, during a period of 28 days and 60 days post study treatment administration, when the patient reached the score of 6, 7 or 8 on the 8-point ordinal scale. | 60 days
All-cause mortality during the period of 28 days and 60 days. | 60 days
Proportion of patients alive and free of respiratory failure, defined as need for IMV, ECMO, noninvasive ventilation, or high-flow nasal cannula oxygen delivery on Days 28 and 60. | 60 days
Cumulative number of vasopressor-free days during the period of 28 days and 60 days. | 60 days
Cumulative number of days in the hospital during the period of 28 days and 60 days. | 60 days
Cumulative number of days in the ICU or Intermediate Care Unit (IMU) during the period of 28 days and 60 days. | 60 days

OTHER OUTCOMES:
Safety - Number and severity of adverse events (AEs) and serious adverse events (SAEs) throughout 60-day follow-up period | 60 days
Safety - Number and severity of AEs and SAEs throughout 180-day follow-up period | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Oren Hershkovitz, PhD, Study Director — Enlivex Therapeutics R&D
Locations (1):
- Hadassah Ein Kerem Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No
Patient data will not contain any information which would make the patient identifiable. Data will be processes and shared using patient study number only.